CLINICAL TRIAL: NCT03990272
Title: Safety and Efficacy of Sublingual Immunotherapy for Allergic Rhinitis Due to Artemisia Annua: a Randomized, Double Blind,Placebo Controlled, Phase III Trial
Brief Title: Safety and Efficacy of Sublingual Immunotherapy for Allergic Rhinitis Due to Artemisia Annua
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Collaborators: Zhejiang Wolwo Bio-Pharmaceutical Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Luo Zhang, vise president of BeijingTongren Hospital, Beijing Tongren Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TR-SLIT-AA-MC
Record Dates: First submitted 2019-06-12; First posted 2019-06-18 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- artemisia annua allergen extract drops (Experimental)
  Interventions: Drug: AIT drops
- Placebo drops (Placebo Comparator)
  Interventions: Drug: placebo drops

INTERVENTIONS:
Drug: AIT drops — once a day
  Arms: artemisia annua allergen extract drops
Drug: placebo drops — once a day
  Arms: Placebo drops

SUMMARY:
Allergic rhinitis (AR) is a common disease of nasal mucosa, affecting 10% to 40% of the population globally. Allergen specific immunotherapy (AIT) is the only etiological treatment available for AR.Traditionally, AIT is divided into subcutaneous immunotherapy (SCIT) and sublingual immunotherapy (SLIT). Artemisia annua is one of the most important allergen that is responsible for seasonal AR in China during July and October.

The trial is a randomized, double-blind, placebo-controlled, multicentred, phase III trial. 702 subjects with allergic rhinitis caused by Artemisia pollen were recruited and randomized to the immunotherapy group and placebo group.

ELIGIBILITY:
Inclusion Criteria:

* presence of seasonal rhinitis symptoms for over 2 years
* artemisia-specific immunoglobulin E (IgE) levels (ImmunoCAP) of class 3 or higher
* patients who have been informed of the nature and aims of the study and have given their written consent, willing to comply with the protocol.
* patients who are able to understand the information given and the consent and complete the daily record card.

Exclusion Criteria:

* patients with severe asthma, perennial allergic rhinitis, cancer or other serious diseases that are unfit to receive allergen immunotherapy
* patients who are taking β-antagonists or have taken systemic corticosteroids in last 4 weeks
* patients whose Humulus- or Artemisiifolia-specific immunoglobulin E (IgE) levels (ImmunoCAP) same as or higher than Artemisia-specific immunoglobulin E (IgE) level.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 702 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-10-22 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
daily combined scores of medication and rhinoconjunctivitis symptoms (CSMRS) | at the peak pollen season(The start was defined as the first of 3 consecutive days with a pollen count of 50 pollen/m3 or greater each day. The end was defined as the last occurrence of 3 consecutive days with ≥50 pollen/m3 each day)
  the daily combined scores of medication and rhinoconjunctivitis symptoms (CSMRS) (ranging from 0 to 6); which was calculated as the combined score of daily average scores of 6 rhinoconjunctivitis symptoms (rhinorrhea, nasal congestion, nasal itching, sneezing, ocular pruritus, and watery eyes) and the daily rescue medication score

SECONDARY OUTCOMES:
daily total nasal symptom score (dTNSS) | at the peak pollen season(The start was defined as the first of 3 consecutive days with a pollen count of 50 pollen/m3 or greater each day. The end was defined as the last occurrence of 3 consecutive days with ≥50 pollen/m3 each day)
  dTNSS was the sum of four nasal symptom scores for nasal congestion, discharge, itching and sneezing (ranging from 0 to 12). Nasal symptoms during the pollen season were rated on a 4-point scale, while 0 = no symptoms, 1 = mild symptoms (sign/symptom clearly present, but minimal awareness; easily tolerated), 2 = moderate symptoms (definite awareness of sign/symptom that is bothersome but tolerable), and 3 = severe symptoms (sign/symptom that is hard to tolerate; causes interference with activities of daily living and/or sleeping)
daily Rescue Medication Scores (dRMS) | at the peak pollen season(The start was defined as the first of 3 consecutive days with a pollen count of 50 pollen/m3 or greater each day. The end was defined as the last occurrence of 3 consecutive days with ≥50 pollen/m3 each day)
  dRMS is the rescue medication score in each day during the peak pollen season (ranging from 0 to 3). 0 = no rescue medication uses, 1 = Oral and/or topical non-sedative H1 antihistamines, 2 = Intranasal corticosteroids (Rhinocort) with/without H1 antihistamines, and 3 = Oral corticosteroids with/without intranasal corticosteroids, with/without H1 antihistamines.
Adverse events | From the first day of SLIT to Visit 9(week 32)
  the occurrence and severity of adverse events (AEs) and the casual relationship between AEs and the experimental drug

CONTACTS AND LOCATIONS:
Locations (13):
- China (13):
  - Beijing Shijitan Hospital, Beijing
  - Beijing Tongren Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - West China Hospital, Sichuan University, Chendu
  - Qingdao Municipal Hospital, Qingdao
  - No. 202 Hospital of PLA （General Hospital of Northern Theater Command ）, Shenyang
  - First Hospital of Shanxi Medical University, Taiyuan
  - Second Hospital of Shanxi Medical University, Taiyuan
  - Tianjin Medical University General Hospital, Tianjin
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi
  - Shaanxi Provincial People's Hospital, Xi'an
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - General Hospital of Ningxia Medical University, Yinchuan